CLINICAL TRIAL: NCT06520852
Title: The Effect of the Use of Artificial Intelligence in the Preparation of Patient Education Material on the Comprehensibility, Actionability and Quality of the Material
Brief Title: The Effect of the Use of Artificial Intelligence in the Preparation of Patient Education Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Associate Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-04/14
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Nursing Education; Artificial Intelligence
MeSH Terms: interventions — Artificial Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group using artificial intelligence tools in addition to traditional tools in preparing educational materials
  Interventions: Other: Group using artificial intelligence tools in addition to traditional tools in preparing educational materials
- Control group (No Intervention): Group using traditional tools in preparing educational materials

INTERVENTIONS:
Other: Group using artificial intelligence tools in addition to traditional tools in preparing educational materials — Students in the intervention group used AI tools in addition to tools such as books, journals, and websites.
  Other Names: artificial intelligence
  Arms: Intervention group

SUMMARY:
This research was conducted to examine the effect of students' use of AI tools while preparing patient education material on the quality, understandability and actionability of the material in terms of content. Students in the control group used auxiliary tools such as books, journals and websites while preparing patient education materials. Students in the intervention group used AI tools in addition to tools such as books, journals, and websites.

DETAILED DESCRIPTION:
This research was conducted to examine the effect of students' use of AI tools while preparing patient education material on the quality, understandability and actionability of the material in terms of content. Students in the control group used auxiliary tools such as books, journals and websites while preparing patient education materials. Students in the intervention group used AI tools in addition to tools such as books, journals, and websites. Patient Education Materials Assessment Tool and Global Quality Scale were used to evaluate the educational materials.

ELIGIBILITY:
Inclusion Criteria:

* agreeing to participate in the study,
* taking the Fundamentals of Nursing II course for the first time,
* not working as a nurse in a hospital or any health institution.

Exclusion Criteria:

* not agreeing to participate in the study
* having prepared patient education materials before
* repeating the Fundamentals of Nursing II course
* not having internet access
* not having a computer or smartphone.

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Understandability of the material | After the students have completed the materials (5 days later)
  Patient Education Materials Assessment Tool for Printable Materials: The tool consists of a total of 26 items, 19 items evaluating the understandability of the materials and 7 items evaluating their actionability. PEMAT scores materials from 0 to 100 points for understandability and actionability.
Actionability of the material | After the students have completed the materials (5 days later)
  Patient Education Materials Assessment Tool for Printable Materials: The tool consists of a total of 26 items, 19 items evaluating the understandability of the materials and 7 items evaluating their actionability. PEMAT scores materials from 0 to 100 points for understandability and actionability.
Quality of the material | After the students have completed the materials (5 days later)
  Global Quality Scale : According to this scale, the quality of the training materials was evaluated on a 5-point scale (1: poor quality, 2: low quality - limited use, 3: somewhat useful, 4: useful, 5: useful-excellent quality).

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA KORKUT, Principal Investigator — TC Erciyes University
Locations (1):
- Sevda Korkut, Talas, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No